CLINICAL TRIAL: NCT03264729
Title: The Acute Effect of Isotonic Versus Isometric Exercise Versus Walking on Pain in Individuals With Plantar Fasciopathy: a Randomised, Participant-blinded, Cross-over Trial
Brief Title: The Acute Effect of Isotonic Versus Isometric Exercise Versus Walking on Pain in Individuals With Plantar Fasciopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Henrik Riel, PhD Student, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N-20170021
Record Dates: First submitted 2017-08-15; First posted 2017-08-29 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Plantar Fasciopathy
Keywords: plantar heel pain
MeSH Terms: interventions — Exercise; Walking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isometric exercise (Experimental)
  Interventions: Other: Isometric exercise
- Isotonic exercise (Active Comparator)
  Interventions: Other: Isotonic exercise
- Walking (Active Comparator)
  Interventions: Other: Walking

INTERVENTIONS:
Other: Isometric exercise — The isometric exercise is performed standing with the forefoot on a step. The participant is instructed to stand still with the ankle joint in neutral and hold this position. Supporting oneself for balance by placing the hands on a wall or a rail is allowed. The participant performs 5 sets of 45-second isometric holds. The load used is the heaviest possible load that the participant is able to withstand for 1 minute. As with the isotonic exercise, if the participant's body weight is inadequate the participant is fitted with a backpack with books and/or weights.
  Arms: Isometric exercise
Other: Isotonic exercise — The isotonic exercise is performed standing with the forefoot on a step. The toes are maximally dorsi-flexed by placing a towel underneath them. The participant is instructed to perform a heel-raise to a maximal plantar flexion in the ankle joint, and afterwards to lower the heel to maximal dorsi flexion. Supporting oneself for balance by placing the hands on a wall or a rail is allowed. The participant performs 4 sets of 8 repetitions with a load of 8RM. The contraction time is 3s concentric, 2s isometric and 3s eccentric and will be guided by a metronome.
  If the participant's body weight is inadequate to reach sufficient loading during the exercises the participant is fitted with a backpack with books and/or weights.
  Arms: Isotonic exercise
Other: Walking — The walking will be performed barefoot and the participant will be instructed in walking at a pace similar to the pace they would use when walking around in their home. The duration of the walking session will be four minutes to match the duration during the exercises.
  Arms: Walking

SUMMARY:
This study investigates the acute effect of isotonic versus isometric exercise versus walking on pain in individuals with plantar heel pain and an ultrasound-diagnosed plantar fasciopathy. The hypothesis is that isometric exercise will induce greater participant rated pain relief than isotonic exercise and walking during aggravating activity.

DETAILED DESCRIPTION:
Participants will be required to attend three sessions (isometric, isotonic, or walking) within a maximum of two weeks. The order in which the participant completes the sessions will be randomised.There will be a minimum of 48 hours between sessions. To account for potential time of day differences in terms of pain, all sessions will be performed within ±1 hour (e.g. if the first session is performed at 10 AM the remaining two sessions will be performed between 9 and 11 AM). After diagnosis, randomisation of the order of which the sessions will be performed, and have their pain during an aggravating activity examined (aggravating activities will be static stance, half squat or heel raise). Subsequently the participants will be instructed in performing either isotonic or isometric heel raise or walking, (determined according to the randomisation) by a physiotherapist.

All statistical analyses will be performed according to a pre-established analysis plan using STATA ver. 14. The assumption of negligible carryover effects is investigated with a preliminary test. The primary analysis will test the presence of a difference in EIH between isotonic and isometric exercise and walking and a 3 X 2 repeated measures ANOVA will be performed. Independent factors will be exercise type (isometric vs. isotonic vs. walking) and time (pre vs. post). If an interaction is found, post-hoc paired t-tests will be performed. The standardised mean difference (effect size) and its confidence intervals will be calculated and presented in a forest plot. Apriori it has been determined that no conclusions will be made favouring either of the exercises nor walking if pain is reduced less than the clinically important difference of 19 mm VAS. In addition, the proportion of clinically relevant pain reductions (i.e. a pain reduction of at least 19 mm VAS) will be calculated. EIH by pain experienced during the aggravating activity before the exercises and walking will also be presented in a plot.

Secondary analyses using a 3 X 2 repeated measures ANOVAs will test if there is a difference in the thickness of the plantar fascia and a difference in PPTs from before to after either of the exercises or walking and a difference in pain experienced during the exercises or walking. If interactions are found post-hoc paired t-tests will be performed. A paired t-test will be performed to investigate potential differences in plantar fascia thickness from before to after the initial PPT and pain aggravating activity are performed. Effect sizes will be calculated for the difference in pressure pain threshold and plantar fascia thickness. The association between thickness of the plantar fascia and the difference in pain from before to after the exercise activities will be investigated using Pearson's correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* History of inferior heel pain for at least three months before enrolment
* Pain on palpation of the medial calcaneal tubercle or the proximal plantar fascia
* Thickness of the plantar fascia of 4.0 mm or greater
* Pain during at least one of three pain aggravating activities (static stance, half squat and heel raise)
* Mean heel pain of ≥ 20 mm on a 100 mm VAS [0mm = no pain, 100mm = worst pain imaginable] during the past week

Exclusion Criteria:

* Below 18 years of age
* History of inflammatory systemic diseases
* Pain or stiffness in the 1st metatarsophalangeal joint to an extent where the exercises cannot be performed
* Prior heel surgery
* Pregnancy
* Pain medication
* Corticosteroid injection for plantar fasciopathy within the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Change in pain | Immediately before and after each exercise/walking
  This is measured during an aggravating task on a 100 mm VAS, where 0 mm is no pain and 100 mm is worst pain imaginable and is also referred to as exercise-induced hypoalgesia (EIH)

SECONDARY OUTCOMES:
Change in pressure pain threshold | Immediately before and after each exercise/walking
  Measured on the tenderest spot under the heel by an algometer in kPa
Change in thickness of the plantar fascia | Immediately before and after each exercise/walking
  Measured by ultrasonography in mm
Pain | During each exercise/walking
  Measured on a 100 mm VAS, where 0 mm is no pain and 100 mm is worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Riel, M.Sc., Principal Investigator — Research Unit for General Practice in Aalborg, Department of Clinical Medicine, Aalborg University
Locations (1):
- Research Unit for General Practice, Aalborg East, Denmark

REFERENCES:
- [Derived] Riel H, Vicenzino B, Jensen MB, Olesen JL, Holden S, Rathleff MS. The effect of isometric exercise on pain in individuals with plantar fasciopathy: A randomized crossover trial. Scand J Med Sci Sports. 2018 Dec;28(12):2643-2650. doi: 10.1111/sms.13296. Epub 2018 Oct 1. PMID 30203866